CLINICAL TRIAL: NCT02550041
Title: Analysis T Cells Response for Identification of Aspergillus Bronchitis With Cystic Fibrosis Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties for inclusions
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UF 9582
Record Dates: First submitted 2015-08-20; First posted 2015-09-15 (Estimated); Last update posted 2019-05-09 (Actual); Status verified 2016-12

CONDITIONS: Cystic Fibrosis Patient; Patient Without Treatment Against A.Fumigatus
Keywords: Bronchitis aspergillus; cystic fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cystic fibrosis (Other)
  Interventions: Other: T specific response for diagnostic of aspergillus bronchitis

INTERVENTIONS:
Other: T specific response for diagnostic of aspergillus bronchitis

SUMMARY:
The study aims to asses the ability of cell tests based on the analysis of the anti-Aspergillus cell responses and identify Aspergillus bronchitis with patients with cystic fibrosis.

In addition, the study will evaluate the contribution of biological classification of aspergillosis according to criteria recently proposed by Baxter et al. compared to the classification used in clinical practice in the hospital of Montpellier.

ELIGIBILITY:
Inclusion Criteria:

* Patient with cystic fibrosis followed at Resource Centers and Cystic Fibrosis Skills (CRCM) Montpellier
* Patient aged 15 or over
* Patient able to understand the nature, purpose and methodology of the study.
* Patient and his legal representative for minors who have given their free and informed consent
* Affiliate or beneficiary of a social security scheme.

Exclusion Criteria:

* Patients on antifungal treatment at the time of sampling
* Pregnant or breastfeeding
* Major protected by law (guardianship, curator or under Backup Justice)
* Inability to understand the nature and goals of the study and / or communication difficulties with the investigator
* Subject attending another search including a period of exclusion still going to run-in

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2015-09-07 (Actual); Primary Completion 2016-09-07 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Number of CD4 T cell response against Aspergillus fumigatus in patients with cystis fibrosis | 12 months
  Analysis T cells response for identification of aspergillus bronchitis with cystic fibrosis patients
Cytokine level of TCD8 | 12 months
  Qualitative Evaluation of cytokine level (IFNg, TNFa, IL10 and IL4) of TCD8 to identify ABPA and aspergillus bronchitis
Cytokine level CD4 cells | 12 months
  Qualitative Evaluation of cytokine level CD4 cells in order to identify ABPA and aspergillus bronchitis

SECONDARY OUTCOMES:
Level of fumigatus specific IgE | 12 months
  Contribution of several biological tests improve classification of aspergillus bronchitis
Level of fumigatus specific IgG | 12 months
  Contribution of several biological tests improve classification of aspergillus bronchitis
Real-time PCR for aspergillus in sputum | 12 months
  Contribution of several biological tests improve classification of aspergillus bronchitis
Galactomannan by enzyme immune assay detection in sputum | 12 months
  Contribution of several biological tests improve classification of aspergillus bronchitis
Levels of cytokine (IFNg, IL10, IL4 and TNF) evaluated by flow cytometry | 12 months
  Contribution of several biological tests improve classification of aspergillus bronchitis
Level of IL10 evaluated by Elispot dedicated to anti-aspergillus CD4 T cells | 12 months
  Contribution of several biological tests improve classification of aspergillus bronchitis
Flow cytometry techniques dedicated to anti-aspergillus CD4 T cell assessment | 12 months
Level of IFNg evaluated by Elispot dedicated to anti-aspergillus CD4 T cells | 12 months
  Contribution of several biological tests improve classification of aspergillus bronchitis
Elispot dedicated to anti-aspergillus CD4 T cell | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Irmb/U1058, Montpellier, France